CLINICAL TRIAL: NCT03728010
Title: Tidal Volume and PEEP Titration in One-Lung Ventilation With Electrical Impedance Tomography
Brief Title: Electrical Impedance Tomography in One-Lung Ventilation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Roberto Gonzalez Cornejo, Anesthesiologist, University of Chile
Other Study IDs: EITOLV001
Record Dates: First submitted 2018-10-09; First posted 2018-11-01 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Ventilator Lung
Keywords: Electrical impedance tomography; One-lung ventilation; Protective ventilation; Ventilator- Induce Lung injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One-Lung Ventilarion: Thoracic surgery cases with one-lung ventilation strategy.
  Interventions: Diagnostic Test: Electrical impedance tomography. Pulmonary mechanics measurement.Arterial gas measurement. Esophageal pressure measurement

INTERVENTIONS:
Diagnostic Test: Electrical impedance tomography. Pulmonary mechanics measurement.Arterial gas measurement. Esophageal pressure measurement — After general anesthesia, patients will be ventilated with three tidal volume level (4, 6 and 8 cc / Kg / IBW), in two levels of PEEP, 6 cm2 H20, and best PEEP, the latter obtained after a recruitment maneuver and decremental titration.

SUMMARY:
Mechanical ventilation can cause damage to the lung parenchyma, this is known as ventilatory induce lung injury (VILI).To avoid this damage, ventilatory strategies have been created, focused on the reduction of tidal volume, airway pressures and use of PEEP (positive end-expiratory pressure), which together are called "protective ventilation".

Although ventilation with protective parameters seems to reduce VILI in one-lung ventilation, the optimal parameters are not clear.

DETAILED DESCRIPTION:
This research aims to describe the ventilation, perfusion and pulmonary mechanics on one-lung ventilation with different levels of tidal volume and PEEP.

An extreme situation of VILI occurs in thoracic surgery, where the atelectasis of a lung is required, ventilating throughout the surgery only the contralateral one. This generates an inflammatory state, with the release of alveolar cytokines from both the non-ventilated and ventilated lungs, which potentiates the development of damage in the lung parenchyma. In addition, one lung ventilation has traditionally been performed with high tidal volume (Vt) values and low PEEP. In this context, the development of VILI is even more probable, so extreme measures of protection in this kind of ventilation are necessary.

The electrical impedance tomography will allow the investigators to obtain a visual and quantitative representation of the areas of ventilation and perfusion of the lung. By relating the tidal volume and PEEP with the tomographic results, it is expected to define mechanical ventilation parameters that achieve the best ventilation/perfusion ratio for patients in one-lung ventilation. Specifically, analyze the distribution and deformation of the ventilated areas in the different lung regions and its correlation with respiratory mechanics and volumetric capnography. This will allow the investigators to make a better definition of the tidal volume and PEEP in patients undergoing one-lung ventilation.

.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) classification I-III
* Age 18-75 Years
* Elective thoracic surgery
* One-Lung Ventilation
* Healthy non ventilated lung

Exclusion Criteria:

* ASA classification > III
* BMI (Body mass index) > 30
* Emergency surgery
* Pregnancy
* Patients includes in other protocols

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients between 18 and 75 years old. With pulmonary diseases that require thoracic surgery with one-lung ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-12-07 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Ventilation/ perfusion ratio | 1 hour
  Electrical impedance tomography.
Pulmonary mechanics | 1 hour
  Airway pressure ,esophageal pressure measurement.
Arterial gas measurement | 20 minutes
  5 samples per patient

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chile Clinical Hospital, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gattinoni L, Protti A, Caironi P, Carlesso E. Ventilator-induced lung injury: the anatomical and physiological framework. Crit Care Med. 2010 Oct;38(10 Suppl):S539-48. doi: 10.1097/CCM.0b013e3181f1fcf7. PMID 21164395
- [Background] Pinhu L, Whitehead T, Evans T, Griffiths M. Ventilator-associated lung injury. Lancet. 2003 Jan 25;361(9354):332-40. doi: 10.1016/S0140-6736(03)12329-X. PMID 12559881
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Futier E, Constantin JM, Paugam-Burtz C, Pascal J, Eurin M, Neuschwander A, Marret E, Beaussier M, Gutton C, Lefrant JY, Allaouchiche B, Verzilli D, Leone M, De Jong A, Bazin JE, Pereira B, Jaber S; IMPROVE Study Group. A trial of intraoperative low-tidal-volume ventilation in abdominal surgery. N Engl J Med. 2013 Aug 1;369(5):428-37. doi: 10.1056/NEJMoa1301082. PMID 23902482
- [Background] El Tahan MR, Pasin L, Marczin N, Landoni G. Impact of Low Tidal Volumes During One-Lung Ventilation. A Meta-Analysis of Randomized Controlled Trials. J Cardiothorac Vasc Anesth. 2017 Oct;31(5):1767-1773. doi: 10.1053/j.jvca.2017.06.015. Epub 2017 Jun 7. PMID 28843606